CLINICAL TRIAL: NCT05379192
Title: How Does Circadian Rhythm Affect Postoperative Pain After Pediatric Acute Appendicit Operation?
Brief Title: The Effect of Circadian Rhytm on Postoperative Pain Undergoing Pediatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Faruk Cicekci (Other)
Responsible Party: Sponsor-Investigator, Faruk Cicekci, Associate Prof., Selcuk University
Organization: Selcuk University (Other)
Other Study IDs: farukcicekci5
Record Dates: First submitted 2022-04-29; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Circadian Rhythm; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Sociodemographic and clinical data of the patients who will be operated between 01:01-07:00 AM will be recorded. The total amount of antiemetic, the time of first antiemetic use, and the VAS scores at the postoperative 1, 2, 3, 6, 9, 12, 15, 18, 21 and 24th hours will also be recorded.
  Interventions: Other: Group 1, Group 2, Group 3, Group 4
- Group 2: Patients who were operated between 07:01-13:00. Sociodemographic and clinical data of the patients who will be operated between 07:00 AM- 01:00 PM will be recorded. The total amount of antiemetic, the time of first antiemetic use, and the VAS scores at the postoperative 1, 2, 3, 6, 9, 12, 15, 18, 21 and 24th hours will also be recorded.
  Interventions: Other: Group 1, Group 2, Group 3, Group 4
- Group 3: Sociodemographic and clinical data of the patients who will be operated between 01:00 - 08:00 PM will be recorded. The total amount of antiemetic, the time of first antiemetic use and the VAS scores at the postoperative 1, 2, 3, 6, 9, 12, 15, 18, 21 and 24th hours will also be recorded.
  Interventions: Other: Group 1, Group 2, Group 3, Group 4
- Group 4: Sociodemographic and clinical data of the patients who will be operated between 08:00 PM -01:00 AM will be recorded. The total amount of antiemetic,the time of first antiemetic use, and the VAS scores at the postoperative 1, 2, 3, 6, 9, 12, 15, 18, 21 and 24th hours will also be recorded.
  Interventions: Other: Group 1, Group 2, Group 3, Group 4

INTERVENTIONS:
Other: Group 1, Group 2, Group 3, Group 4 — The total amount of antiemetic,the time of first antiemetic use and VAS scores at 1, 2, 3, 6, 9, 12, 15, 18, 21 and 24th hours postoperatively will also be recorded according to circadian rhythm

SUMMARY:
These circadian rhythms are self-sustained, endogenous oscillations generated by circadian clocks that persist with a period of around 24 -h under constant conditions. Multiple clinical and foundational science studies report that circadian rhythm disruption can directly alter pain thresholds. Altered circadian pain rhythms manifest inconsistently in various disease states. circadian differences exist in tolerability of administration as well as in effectiveness of analgesia during surgical, obstetric, and dental procedures, with the majority of studies demonstrating highest pain sensitivity during the overnight or early morning hours. Although the relationship between pain states and circadian rhythm has been studied in various surgical procedures and chronic pain syndromes, there is little literature examining the relationship between postoperative pain and circadian rhythm in pediatric surgical procedures. Therefore, it was aimed to evaluate the relationship between postoperative pain and circadian rhythm after pediatric acute appendicitis surgery.

DETAILED DESCRIPTION:
This study will be conducted with the data to be obtained from the Anesthesiology Surgery Form and Pediatric Surgery Service Forms in 200 patients aged 6-18 years, after the approval of the Faculty Local Ethics Committee in the Department of Anesthesiology, Faculty of Medicine, Selcuk University. According to the time the patients were taken into the operation, Group 1; 01:01-07:00, Group 2; 07:01-13:00, Group 3; 13:01-20:00 and Group 4; 20:01-01:00, It will be divided into four groups between. The files of the patients will be examined and demographic data such as age (year), body weight (kg), height (cm), gender, ASA scores (I-III), anesthesia and surgery time, anesthesia and surgery time will be recorded. Intraoperative vital signs; systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP), heart rate (HR) oxygen saturation (SpO2) Endtidal CO2 and temperature before operation (control) and 5, 10, 15, 20, 25 and 30 minutes (min) and at the end of the process (end) data will also be saved. Perioperative side effects such as nausea-vomiting, hypotension, bradycardia, tremor, respiratory distress, sore throat, headache, and dizziness symptoms will be noted if they occur. The routinely applied analgesic protocol and vital signs in the postoperative pediatric surgery service, the total amount of analgesic administered, the time to first analgesia requirement and VAS scores at 1, 2, 3, 6, 9, 12, 15, 18, 21 and 24th hours will also be recorded. There will be no interference with the routinely applied analgesic protocol.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical condition I-II,
* Undergoing acute appendicitis,
* Patients aged 6-18 years

Exclusion Criteria:

* ASA ≥ III,
* Uncontrolled chronic, metabolic disease,
* Opioid or analgesic use in the last 10 days,
* Acute peritonitis or sepsis
* History of abnormal operation or recovery from anesthesia,
* Patients with parents who are unwilling to give informed consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Postoperative pain differs in both sexes according to the circadian rhythm.
Study Population: Pediatric patient population of both sexes aged 6-18 years
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The postoperative VAS pain scores | 1st hours , postoperatively
  The VAS scores at 1st will be recorded.
The postoperative VAS pain scores | 2nd hours , postoperatively
  The VAS scores at 2nd will be recorded.
The postoperative VAS pain scores | 3th hours , postoperatively
  The VAS scores at 3th will be recorded.
The postoperative VAS pain scores | 6th hours , postoperatively
  The VAS scores at 6th will be recorded.
The postoperative VAS pain scores | 9th hours , postoperatively
  The VAS scores at 9th will be recorded.
The postoperative VAS pain scores | 12th hours , postoperatively
  The VAS scores at 12th will be recorded.
The postoperative VAS pain scores | 15th hours , postoperatively
  The VAS scores at 15th will be recorded.
The postoperative VAS pain scores | 18th hours , postoperatively
  The VAS scores at 18th will be recorded.
The postoperative VAS pain scores | 21th hours , postoperatively
  The VAS scores at 21th will be recorded.
The postoperative VAS pain scores | 24th hours , postoperatively
  The VAS scores at 24th will be recorded.

SECONDARY OUTCOMES:
The total amount of analgesic | 24 hours, postoperatively
  The total amount of analgesic will be recorded postoperativly .
the time to first analgesia requirement | 24 hours, postoperatively
  the time to first analgesia requirement will be recorded postoperativly .

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, School of Medicine, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not have a plan to make individual participant data (IPD) available to other researchers.